CLINICAL TRIAL: NCT00085501
Title: Phase II Selection Design Trial Of Concurrent Chemotherapy + Cetuximab Vs. Chemotherapy Followed By Cetuximab In Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: S0342: Paclitaxel, Carboplatin, and Cetuximab in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000370806; S0342 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cetuximab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: cetuximab; Drug: carboplatin; Drug: paclitaxel
- 2 (Active Comparator)
  Interventions: Drug: cetuximab; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: cetuximab — Arm 1: 400 mg/m2 (Initial dose), 2 hour IV infusion on Day 1, Week 1 only. 250 mg/m2 (Subsequent doses), 1 hour IV infusion, on Day 1 weekly starting at Week 2.
  Arm 2: 400 mg/m2 (Initial dose), 2 hour IV infusion on Week 13 ONLY 250 mg/m2 (Subsequent doses), 1 hour IV infusion, weekly starting at Week 14.
Drug: carboplatin — Arm 1: AUC=6 30 minute IV infusion immediately following paclitaxel on Day 1 q 21 days x 4 starting at Week 2
  Arm 2: AUC=6 30 minute IV infusion immediately following paclitaxel on Day 1 q 21 days x 4 starting at Week 1
Drug: paclitaxel — Arm 1: 225 mg/m2 3 hour IV infusion 1 hour following cetuximab on Day 1, q 21 days x 4 Starting at Week 4.
  Arm 2: 225 mg/m2 3 hour IV infusion 1 hour following cetuximab on Day 1, q 21 days x 4 Starting at Week 1.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining more than one chemotherapy drug with a monoclonal antibody may kill more tumor cells. It is not yet known whether cetuximab is more effective when given at the same time as chemotherapy or following chemotherapy.

PURPOSE: This randomized phase II trial is studying how well giving cetuximab at the same time as combination chemotherapy works compared to giving cetuximab after combination chemotherapy in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with selected stage IIIB or stage IV non-small cell lung cancer treated with concurrent vs sequential paclitaxel, carboplatin, and cetuximab.

Secondary

* Compare response rates (confirmed and unconfirmed, complete and partial) in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Correlate epidermal growth factor receptor polymorphisms and downstream biomarkers with response to cetuximab in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (concurrent cetuximab): Patients receive cetuximab IV over 1 hour (over 2 hours on day 1 of course 1 only) on days 1, 8, and 15 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 8. Treatment repeats every 21 days for a total of 4 courses (12 weeks) in the absence of disease progression or unacceptable toxicity. Beginning on week 13, patients receive single-agent cetuximab IV over 1 hour once weekly in the absence of disease progression or unacceptable toxicity.
* Arm II (sequential cetuximab): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for a total of 4 courses (12 weeks) in the absence of disease progression or unacceptable toxicity. Beginning on week 13, patients receive single-agent cetuximab IV over 1 hour (over 2 hours on week 13 only) once weekly in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 180 patients (90 per treatment arm) will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) of one of the following stages:

  * Newly diagnosed selected stage IIIB disease (T4 lesion due to malignant pleural effusion, any N, M0)
  * Newly diagnosed stage IV disease (any T, any N, M1)
  * Recurrent stage IV disease after prior surgery or radiotherapy
* The following subtypes are eligible:

  * Adenocarcinoma
  * Squamous cell carcinoma
  * Large cell carcinoma
  * Unspecified
* Measurable disease by CT scan, MRI, x-ray, or physical exam

  * Pleural effusions, ascites, or laboratory parameters are not acceptable as the only evidence of disease
  * Not within prior radiotherapy field unless a new lesion is present
  * Not within area of prior surgical resection
* No known brain metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 mg/dL

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT or SGPT ≤ 2 times ULN
* Alkaline phosphatase ≤ 2 times ULN
* No known acute hepatitis

Renal

* Creatinine ≤ ULN
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No significant cardiac disease
* No uncontrolled hypertension
* No unstable angina
* No congestive heart failure

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* No active or uncontrolled infection
* No sensory neuropathy ≥ grade 2
* No known human anti-mouse antibodies
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for NSCLC
* No prior chimeric or murine monoclonal antibody therapy
* No prior cetuximab

Chemotherapy

* No prior systemic chemotherapy for NSCLC

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered

Surgery

* See Disease Characteristics
* At least 2 weeks since prior thoracic or major surgery and recovered

Other

* No prior gefitinib or other investigational agents that target the epidermal growth factor receptor pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2004-07; Primary Completion 2007-08 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Select a regimen based on overall survival | From date of registration until the date of progression or date of death from any cause, whichever came first, assessed up to 3 years
  To select a regimen based on overall survival via a Phase II selection design of chemotherapy in conjunction with cetuximab (concurrent vs. sequential) for Phase III testing against chemotherapy alone in Stage IIIB and Stage IV non-small cell lung cancer.
Response rate (confirmed and unconfirmed, complete and partial response) | From date of registration until the date of progression or date of death from any cause, whichever came first, assessed up to 3 years
  To evaluate response rates (confirmed and unconfirmed, complete and partial) of patients with selected Stage IIIB and Stage IV NSCLC treated with paclitaxel and carboplatin with concurrent cetuximab or paclitaxel and carboplatin followed by cetuximab.
Toxicities | From date of registration until the date of progression or date of death from any cause, whichever came first, assessed up to 3 years
  To evaluate the toxicities of the two treatment regimens in patients with selected Stage IIIB and Stage IV NSCLC.

SECONDARY OUTCOMES:
Correlation of epidermal growth factor receptor polymorphisms and downstream biomarkers with response | At prestudy
  To conduct exploratory molecular correlative studies of the EGFR-HER signaling pathways examining activated phosphoproteins, oncogenic mutations and rates of proliferation and apoptosis in patient tissues (see S9925 for details).
Evaluate EGFR polymorphisms | At prestudy and week 5
  To evaluate EGFR polymorphisms as a potential correlate for response to cetuximab (see S9925 for details).

CONTACTS AND LOCATIONS:
Overall Officials: Roy S. Herbst, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center; Karen Kelly, MD, Principal Investigator — University of Colorado, Denver; David R. Gandara, MD, Principal Investigator — University of California, Davis
Locations (163):
- United States (163):
  - Alaska Regional Hospital, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Valley Memorial Hospital, Livermore, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Highland General Hospital, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - CCOP - Santa Rosa Memorial Hospital, Sana Rosa, California
  - St. Anthony Central Hospital, Denver, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - St. Anthony North Hospital, Westminster, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Piedmont Hospital, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Augusta Oncology Associates, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Hematology Oncology Consultants Ltd., Naperville, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Tulane Cancer Center, New Orleans, Louisiana
  - Cancer Treatment Center at Christus Schumpert St. Mary Place, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cancer Care Center at Battle Creek Health System, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Spectrum Health Hospital - Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Mount Clemens General Hospital, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Hospital, Pontiac, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Kessler Air Force Base, Mississippi
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Adirondack Cancer Care, Glens Falls, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Tri-Health Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - St. Charles Medical Center, Bend, Oregon
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Comprehensive Cancer Center at Legacy Good Samaritan Hospital & Medical Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Salem Hospital Regional Cancer Center, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Arlington Cancer Center - Arlington, Arlington, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Cancer Care Center at Skagit Valley Hospital, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - North Star Lodge Cancer Center, Yakima, Washington
  - Washington Hematology - Oncology Specialists, Yakima, Washington

REFERENCES:
- [Background] Franklin WA, Gandara DR, Kim ES, et al.: SWOG S0342 and S0536: expression of EGFR protein and markers of epithelial-mesenchymal transformation (EMT) in cetuximab/chemotherapy-treated non-small cell lung cancer (NSCLC). [Abstract] J Clin Oncol 27 (Suppl 15): A-11076, 2009.
- [Background] Mack PC, Holland WS, Redman M, et al.: KRAS mutation analysis in cetuximab-treated advanced stage non-small cell lung cancer (NSCLC): SWOG experience with S0342 and S0536. [Abstract] J Clin Oncol 27 (Suppl15): A-8022, 2009.
- [Result] Hirsch FR, Herbst RS, Olsen C, Chansky K, Crowley J, Kelly K, Franklin WA, Bunn PA Jr, Varella-Garcia M, Gandara DR. Increased EGFR gene copy number detected by fluorescent in situ hybridization predicts outcome in non-small-cell lung cancer patients treated with cetuximab and chemotherapy. J Clin Oncol. 2008 Jul 10;26(20):3351-7. doi: 10.1200/JCO.2007.14.0111. PMID 18612151
- [Result] Herbst RS, Chansky K, Kelly K, et al.: A phase II randomized selection trial evaluating concurrent chemotherapy plus cetuximab or chemotherapy followed by cetuximab in patients with advanced non-small cell lung cancer (NSCLC): final report of SWOG 0342. [Abstract] J Clin Oncol 25 (Suppl 18): A-7545, 395s, 2007.
- [Result] Kelly K, Herbst RS, Crowley JJ, et al.: Concurrent chemotherapy plus cetuximab or chemotherapy followed by cetuximab in advanced non-small cell lung cancer (NSCLC): a randomized phase II selectional trial SWOG 0342. [Abstract] J Clin Oncol 24 (Suppl 18): A-7015, 367s, 2006.